CLINICAL TRIAL: NCT06264219
Title: "Restoration of the Gut Microbiome After Cesarean Section (RestoreGut)" - a Double-blinded Randomized Controlled Feasibility Trial
Brief Title: Restoration of the Gut Microbiome After Cesarean Section
Acronym: RestoreGut
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Professor Klaus Bønnelykke (Other)
Responsible Party: Sponsor-Investigator, Professor Klaus Bønnelykke, Professor PhD, Head of COPSAC, Copenhagen Studies on Asthma in Childhood
Organization: Copenhagen Studies on Asthma in Childhood (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-24002284
Record Dates: First submitted 2024-02-12; First posted 2024-02-16 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- FMT (Fecal microbiota transplantation) (Active Comparator): Mother-to-infant fecal microbiota transplantation
  Interventions: Biological: Microbiome restoration - FMT
- FVT (Fecal virome transplantation) (Active Comparator): Mother-to-infant fecal virome transplantation
  Interventions: Biological: Microbiome restoration - FVT
- Placebo (Placebo Comparator): Inactive solution buffer placebo
  Interventions: Biological: Placebo
- Vaginal control group (Other): Non-randomized control group used for secondary outcomes comparisons.
  Interventions: Other: Vaginal birth, untreated control

INTERVENTIONS:
Biological: Microbiome restoration - FMT — Pathogen-free microbiota from maternal stool sample is transferred from mother to infant.
  Other Names: Fecal Microbiota Transplantation
  Arms: FMT (Fecal microbiota transplantation)
Biological: Microbiome restoration - FVT — Sterile-filtered and ultracentrifuged FMT, containing only viruses, is transferred from mother to infant.
  Other Names: Fecal Virome Transplantation
  Arms: FVT (Fecal virome transplantation)
Biological: Placebo — Inactive solution buffer
  Arms: Placebo
Other: Vaginal birth, untreated control — No intervention. This group is for secondary outcomes comparisons.
  Arms: Vaginal control group

SUMMARY:
This study aims to develop a therapy for restoring the gut microbiome in infants born via CS. The Study will conduct a randomized, placebo-controlled feasibility trial to assess the ability of microbiome restoration by FMT and FVT in infants born by cesarean section.

DETAILED DESCRIPTION:
When a child is born vaginally, the passage through the birth canal provides the first and very important bacterial colonization. As the child ages, various environmental exposures, such as dietary changes and the presence of older siblings in the home, facilitate a natural maturation of the child's gut microbiome, providing a vast and continuous stimulation of the child's developing immune system. However, factors such as mode of delivery and intrapartum antibiotics can perturb this natural developmental process and cause long-term microbial derangements. The prevalence of cesarean section (CS) birth has increased globally in recent decades, and with it, antibiotic treatment to prevent perinatal infection. Similar patterns have occurred for the prevalence of chronic childhood disease, particularly asthma, with an estimated 300 million asthmatic cases worldwide.

The hypothesis is that early intervention with mother-to-infant FMT can restore a CS-perturbed microbiome to a normal microbial trajectory. Another hypothesis is that seeding the virome fraction (FVT) will cause the neonate's microbiome to resemble the mother's since the transferred phages are enriched and preserved in the intestinal mucus layer, thereby providing the recipient with selective antimicrobial protection while allowing species resembling the mother's own to establish during subsequent bacterial transmission.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < week 38+0 days
* Proficient in spoken/written Danish
* Single pregnancy (no twins or triplets)
* Pre-pregnancy BMI between 18.5 and 35 kg/m2
* No chronic intestinal, endocrine, cardiac, or kidney disorders
* No known gestational complications (gestational diabetes, preeclampsia, gestational hypothyroidism)
* No regular use of prescription medication or any drugs that, in the research team's opinion, may interfere with the study's results.
* Willingness to abstain from giving the child products with probiotics (fermented dairy like yogurt or A38 are allowed).

Exclusion Criteria:

Maternal:

* Use of antibiotics within one month of stool donation
* Acute gastroenteritis within one month of stool donation
* Use of antibiotics within one month of birth
* Time since last travel abroad relative to data of fecal donation according to the requirements for blood donations ("Regler for tappepauser" - blooddonor.dk)
* Positive test results for pathogens during donor material screening.
* Antibiotic treatment at birth (vaginal births only)
* Spontaneous onset of labor or emergency cesarean section before scheduled cesarean section.

Infant:

* Instances of major birth defects or intrauterine growth retardation (IUGR)
* Infants requiring pediatric support at the time of transplant administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 80 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Microbial compositional differences to placebo-treated infants | During the first year of life
  Intestinal microbiome composition, assessed by metagenomic sequencing of fecal matter bacterial DNA, quantified by beta-diversity indices.

SECONDARY OUTCOMES:
Microbial compositional resemblance to vaginally-born infants | During the first year of life
  Intestinal microbiome composition, assessed by metagenomic sequencing of fecal matter bacterial DNA, quantified by beta-diversity indices.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bønnelykke, MD, PhD, Study Chair — Head of COPSAC
Locations (2):
- Denmark (2):
  - Copsac, DBAC, Gentofte Municipality, Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
Individual-level personally identifiable clinical data from the children participating in the cohort cannot be made freely available, to protect the privacy of the participants and their families, in accordance with the Danish Data Protection Act and European Regulation 2016/679 of the European Parliament and of the Council (GDPR) that prohibit distribution even in pseudo-anonymized form. However, research collaborations are welcome, and data can be made available under a joint research collaboration by contacting the COPSAC Data Protection Officer (DPO), Ulrik Ralfkiaer, PhD (dpo@dbac.dk).
Time Frame: Sequences will be deposited in the Sequence Read Archive repository after publication. External research collaborations are welcome after the initial publication.
Access Criteria: Sequences will be openly accessible, individual participant data only under research collaborations.